CLINICAL TRIAL: NCT01977209
Title: A Randomized, Double Blind, Placebo-controlled Multiple-center Phase III Trial of Gossypol Combined With Docetaxel and Cisplatin Scheme in Advanced Non Small-cell Lung Cancers With APE1 High Expression
Brief Title: Gossypol Combined With Docetaxel and Cisplatin Scheme in Advanced Non Small-cell Lung Cancers With APE1 High Expression
Acronym: GTCA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Dong Wang, chief physician, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTCA
Record Dates: First submitted 2013-10-19; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Gossypol; APE1; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gossypol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Docetaxel 75mg/m2/iv over 90min and cisplatin 75mg/m2/iv over 90min on day 1. Gossypol 20mg from day 1 to day 14. repeat Q 3weeks. Four cycles.
  Interventions: Drug: Gossypol
- Arm B (Placebo Comparator): Docetaxel 75mg/m2/iv over 90min and cisplatin 75mg/m2/iv over 90min on day 1. Placebo from day 1 to day 14. repeat Q 3weeks. Four cycles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gossypol
  Arms: Arm A
Drug: Placebo
  Arms: Arm B

SUMMARY:
The investigators' experimental study found that gossypol was the natural inhibitor of apyrimidinic endonuclease 1 (APE1) and clinical study observed that high expression of APE1 was relative to the platinum-resistance in non-small cell lung cancer. Thus the purpose of this study is to find out whether gossypol can improve the sensitivity of cisplatin-based chemotherapy in the non-small cell lung cancer with apurinic apyrimidinic endonuclease 1 (APE1) high expression

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of NSCLC, Stage IIIB/IV.
* Males or females between 18 Years to 75 Years.
* No prior cisplatin-based chemotherapy, if the surgery or radiotherapy has been administered, the interval is at least above four weeks. The interval for targeted therapy such as EGFR TKI is above 2 weeks.
* Performance status of 0, 1 on the ECOG criteria. Expected survival is above three months.
* At least one unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST. 2000).
* Patients can have the brain / meningeal metastasis history, but the metastasis must be treated by operation or radiotherapy), and clinically stable for at least 2 months.
* Adequate hematologic (neutrophil count >= 1,500/uL, platelets >= 100,000/uL), hepatic (transaminase =< upper normal limit(UNL)x2.5, bilirubin level =< UNLx1.5), and renal (creatinine =< UNL) function.
* Patient compliance that allow adequate follow-up. Informed consent from patient or patient's relative.
* APE1 IHC (++ or +++).
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 2 months after trial. If male, use of an approved contraceptive method during the study and 2 months afterwards. Females with childbearing potential must have a urine negative HCG test within 7 days prior to the study enrollment.
* No concomitant prescriptions including cyclosporin A, valproic acid, phenobarbital, phenytoin, ketoconazole.

Exclusion Criteria:

* Inability to comply with protocol or study procedures.
* Medically uncontrolled serious heart, lung, neurological, psychological, metabolic disease.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Pregnant or breast-feeding.
* Enrollment in other study within 30 days.
* Brain metastasis with symptoms.
* Hypokalemic periodic paralysis history.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | the first day of treatment to the date that disease progression is reported; assesed up to 4 years

SECONDARY OUTCOMES:
Overall survival | the first day of treatment to death or last survival confirm date; assesed up to 4 years
Tumor response rate | Up to 4 years
  The ratio between the number of responders and number of patients assessable for tumor response
Toxicity | the first date of treatment to 30 days after the last dose of study drug
  Toxicity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Quality of life | the day before every cycle of chemotherapy; 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wang, PH.D., Principal Investigator — Cancer Center, Daping Hospital, Third Military Medical University
Locations (6):
- China (6):
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Chongqing Zhongshan Hospital, Chongqing, Chongqing Municipality
  - Fuling Central Hospital, Chongqing, Chongqing Municipality
  - Jiangjin Central Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Medical University Of Chongqing, Chongqing, Chongqing Municipality
  - Three Gorges Central Hospital, Chongqing, Chongqing Municipality

REFERENCES:
- [Background] Olaussen KA, Dunant A, Fouret P, Brambilla E, Andre F, Haddad V, Taranchon E, Filipits M, Pirker R, Popper HH, Stahel R, Sabatier L, Pignon JP, Tursz T, Le Chevalier T, Soria JC; IALT Bio Investigators. DNA repair by ERCC1 in non-small-cell lung cancer and cisplatin-based adjuvant chemotherapy. N Engl J Med. 2006 Sep 7;355(10):983-91. doi: 10.1056/NEJMoa060570. PMID 16957145
- [Background] Kelley MR, Georgiadis MM, Fishel ML. APE1/Ref-1 role in redox signaling: translational applications of targeting the redox function of the DNA repair/redox protein APE1/Ref-1. Curr Mol Pharmacol. 2012 Jan;5(1):36-53. doi: 10.2174/1874467211205010036. PMID 22122463
- [Background] Wang D, Xiang DB, Yang XQ, Chen LS, Li MX, Zhong ZY, Zhang YS. APE1 overexpression is associated with cisplatin resistance in non-small cell lung cancer and targeted inhibition of APE1 enhances the activity of cisplatin in A549 cells. Lung Cancer. 2009 Dec;66(3):298-304. doi: 10.1016/j.lungcan.2009.02.019. Epub 2009 Mar 25. PMID 19324449
- [Background] Sonpavde G, Matveev V, Burke JM, Caton JR, Fleming MT, Hutson TE, Galsky MD, Berry WR, Karlov P, Holmlund JT, Wood BA, Brookes M, Leopold L. Randomized phase II trial of docetaxel plus prednisone in combination with placebo or AT-101, an oral small molecule Bcl-2 family antagonist, as first-line therapy for metastatic castration-resistant prostate cancer. Ann Oncol. 2012 Jul;23(7):1803-8. doi: 10.1093/annonc/mdr555. Epub 2011 Nov 23. PMID 22112969
- [Background] Ready N, Karaseva NA, Orlov SV, Luft AV, Popovych O, Holmlund JT, Wood BA, Leopold L. Double-blind, placebo-controlled, randomized phase 2 study of the proapoptotic agent AT-101 plus docetaxel, in second-line non-small cell lung cancer. J Thorac Oncol. 2011 Apr;6(4):781-5. doi: 10.1097/JTO.0b013e31820a0ea6. PMID 21289522
- [Background] Bepler G, Williams C, Schell MJ, Chen W, Zheng Z, Simon G, Gadgeel S, Zhao X, Schreiber F, Brahmer J, Chiappori A, Tanvetyanon T, Pinder-Schenck M, Gray J, Haura E, Antonia S, Fischer JR. Randomized international phase III trial of ERCC1 and RRM1 expression-based chemotherapy versus gemcitabine/carboplatin in advanced non-small-cell lung cancer. J Clin Oncol. 2013 Jul 1;31(19):2404-12. doi: 10.1200/JCO.2012.46.9783. Epub 2013 May 20. PMID 23690416